CLINICAL TRIAL: NCT01027104
Title: Evaluation of a Firearm Injury Prevention Web-based Curriculum
Brief Title: Evaluation of a Resident Curriculum in Firearm Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Leslie M. Dingeldein, Children's Memorial Hospital
Model: Parallel | Masking: None
Other Study IDs: 2008-13313
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Injury; Training
Keywords: injury prevention; firearms; training; counseling; medical education; safety; anticipatory guidance; Firearm injury prevention anticipatory guidance
MeSH Terms: conditions — Wounds and Injuries | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Education — Firearm injury prevention anticipatory guidance curriculum

SUMMARY:
The purpose of this project is to evaluate the efficacy of a web-based curriculum designed to teach pediatric practitioners how to provide injury prevention anticipatory guidance, emphasizing firearm injury prevention in a clinic setting. Data will be collected regarding the curriculum's effectiveness using a web-based questionnaire which will be administered to pediatric residents prior to, immediately post, and six months following completion of the curriculum. Pre- and post-test questionnaires will be compared. Residents will also be asked to evaluate the curriculum by completing a survey. We hypothesize that the curriculum will improve residents' knowledge, attitudes and beliefs, and self-efficacy regarding firearm injury prevention anticipatory guidance.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric resident at Children's Memorial Hospital

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Likert-scale based testing | pre-test, post-test, and 6-months post-test

CONTACTS AND LOCATIONS:
Overall Officials: Leslie M Dingeldein, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Karen Sheehan, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- See also: Link to curriculum used in this study — http://www.injury-ed.org